CLINICAL TRIAL: NCT03940352
Title: A Phase Ib, Multi-arm, Open-label, Study of HDM201 in Combination With MBG453 or Venetoclax in Adult Subjects With Acute Myeloid Leukemia (AML) or High-risk Myelodysplastic Syndrome (MDS)
Brief Title: HDM201 in Combination With MBG453 or Venetoclax in Patients With Acute Myeloid Leukemia (AML) or High-risk Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHDM201H12101C; 2018-004001-62 (EudraCT Number)
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia (AML); High-risk Myelodysplastic Syndrome (MDS)
Keywords: Phase Ib; BHLRM; AML; MDS; HDM201; TP53; MBG453; TIM-3; venetoclax; Bcl-2
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — siremadlin; sabatolimab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- treatment arm1: HDM201+MBG453 (Experimental): Phase Ib (escalation)
  Interventions: Drug: HDM201; Biological: MBG453
- treatment arm2: HDM201+venetoclax (Experimental): Phase Ib (escalation)
  Interventions: Drug: HDM201; Drug: Venetoclax

INTERVENTIONS:
Drug: HDM201 — Capsule
Biological: MBG453 — LIVI (Liquid in vial) Concentrate for Solution for infusion
  Arms: treatment arm1: HDM201+MBG453
Drug: Venetoclax — Tablet
  Arms: treatment arm2: HDM201+venetoclax

SUMMARY:
This was a phase 1b, multi-arm, open-label study of HDM201 in combination with MBG453 or venetoclax in subjects with AML or high-risk MDS.

For all subjects, TP53wt status had to be characterized by, at a minimum, no mutations noted in exons 5, 6, 7 and 8.

Two treatment arms enrolled subjects in parallel to characterize the safety, tolerability, PK, PD and preliminary antitumor activity of HDM201+MBG453 (treatment arm 1) and HDM201+venetoclax (treatment arm 2).

* In the treatment arm 1, subjects received HDM201 in combination with MBG453.
* In the treatment arm 2, subjects received HDM201 in combination with venetoclax. Venetoclax dose was gradually increased (ramp-up) over a period of 4 to 5 days to achieve the daily target dose tested that was subsequently continued.

Upon the completion of the escalation part, MTD(s) and/or RD(s) of HDM201 in combination with MBG453 or venetoclax in AML and high-risk MDS subjects was planned to be determined for each treatment arm.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patients ≥ 18 years of age at the date of ICF signature who present with one of the following:

  1. Relapsed/refractory AML following ≥1 prior therapies (but ≤3 prior therapies) who have relapsed or exhibited refractory disease (primary failure) and are deemed by the Investigator not to be candidates for standard therapy, including re-induction with cytarabine or other established chemotherapy regimens for patients with AML (patients who are suitable for standard re-induction chemotherapy or hematopoietic stem cell transplantation and willing to receive it are excluded)
  2. First line AML patient unfit for standard induction chemotherapy (includes both de novo and secondary AML), except in countries where approved therapies are available. Patients who are suitable for hematopoietic stem cell transplantation and willing to receive it are excluded.
  3. High-risk MDS patient (high and very high-risk groups according to rIPSS) who have failed hypomethylating agent therapy.
* ECOG performance status ≤ 1
* TP53wt tumor. At minimum exons 5, 6, 7 and 8 in the TP53 gene must be sequenced and determined to contain no mutations. The TP53 status must be obtained from a bone-marrow sample, collected no longer than 3 months before signing the main ICF.
* Patient must be a candidate for serial bone marrow aspirate and/or biopsy according to the institutional guidelines and be willing to undergo a bone marrow aspirate and/or biopsy at screening, during and at the end of therapy on this study. Exceptions may be considered after documented discussion with Novartis.

Main Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

* Prior combination treatment with compounds having the same mode of action:

  * mdm2 or mdm4 inhibitors combined with TIM-3 inhibitors (for patients enrolled in treatment arm1)
  * mdm2 or mdm4 inhibitors combined with Bcl-2 inhibitor (for patients enrolled in treatment arm2)
* History of severe hypersensitivity reactions to any ingredient of study drug(s) and other monoclonal antibodies (mAbs) and/or their excipients.
* Patients with acute promyelocytic leukemia with PML-RARA.
* Allogeneic stem cell transplant (HSCT) within last 6 months and/or active GvHD requiring systemic immunosuppressive therapy.
* GI disorders impacting absorption of oral HDM201 or venetoclax.
* Evidence of active bleeding or bleeding diathesis or major coagulopathy (including familial).
* Patients with active, known or suspected autoimmune disease (treatment arm 1 only).

Other eligibility criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) as a measure of safety | at month 24
  Month 24 is assumed to be study end
Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) as a measure of safety | at month 24
  Month 24 is assumed to be study end
Incidence of dose limiting toxicities (DLTs) of treatment | at day 28
  end of first cycle
Frequency of dose interuptions | at month 24
  Month 24 is assumed to be study end
Frequency of dose reductions | at month 24
  Month 24 is assumed to be study end
Dose intensities | at month 24
  measured in mg/ day Month 24 is assumed to be study end

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | at month 24
  Month 24 is assumed to be study end
Best Overall Response (BOR) | at month 24
  Month 24 is assumed to be study end
Event Free Survival (EFS) for AML (Cheson 2003) or Progression Free Survival (PFS) for MDS (Cheson 2006) | at month 24
  Month 24 is assumed to be study end
Relapse Free Survival (RFS) for AML (Cheson 2003) or Time To Response (TTR) for MDS (Cheson 2006) | at month 24
  Month 24 is assumed to be study end
Duration Of Response (DOR) for AML (Cheson 2003) and MDS (Cheson 2006) | at month 24
  Month 24 is assumed to be study end
Presence of anti-MBG453 antibodies (treatment arm 1 HD201+MBG453) | at Day 1, Day 29 and at month 24
Concentration of HDM201 (Treatment arm 1 HDM201+MBG453 and treatment arm 2 HDM201+venetoclax) | at Day 1, Day 2, Day 5, Day 6 and Day 29
Concentration of MBG453 (treatment arm 1 HDM201+MBG453) | at Day 1, Day 2, Day 8, Day 11, Day 15, Day 29 and at month 24
Concentration of venetoclax (treatment arm 2 HDM201+venetoclax) | at Day 1, Day 2, Day 3, Day 5, Day 6, Day 8, Day 9, Day 14, Day 15 and Day 29
PK parameter (AUC) of HDM201 (Treatment arm 1 HDM201+MBG453 and treatment arm 2 HDM201+venetoclax) | at month 6
  Cycle 6
PK parameter (Cmax) of HDM201 (Treatment arm 1 HDM201+MBG453 and treatment arm 2 HDM201+venetoclax) | at month 6
  Cycle 6
PK parameter (Tmax) of HDM201 (Treatment arm 1 HDM201+MBG453 and treatment arm 2 HDM201+venetoclax) | at month 6
  Cycle 6
PK parameter (AUC) of MBG453 (treatment arm 1 HDM201+MBG453) | at month 6
  Cycle 6
PK parameter (Cmax) of MBG453 (treatment arm 1 HDM201+MBG453) | at month 6
  Cycle 6
PK parameter (Tmax) of MBG453 (treatment arm 1 HDM201+MBG453) | at month 6
  Cycle 6
PK parameter (AUC) of venetoclax (treatment arm 2 HDM201+venetoclax) | at month 6
  Cycle 6
PK parameter (Cmax) of venetoclax (treatment arm 2 HDM201+venetoclax) | at month 6
  Cycle 6
PK parameter (Tmax) of venetoclax (treatment arm 2 HDM201+venetoclax) | at month 6
  Cycle 6
Changes from baseline in GDF-15 (Treatment arm 1 HDM201+MBG453 and treatment arm 2 HDM201+venetoclax) | at Day 1 and Day 2
Changes from baseline in soluble TIM-3 (Treatment arm 1 HDM201+MBG453) | at month 6
  Cycle 6

CONTACTS AND LOCATIONS:
Locations (9):
- Duke University Medical Center ., Durham, North Carolina, United States
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Helsinki, Finland
- Germany (2):
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Würzburg
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18331
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2783